CLINICAL TRIAL: NCT00934505
Title: Predictive Value of FDG-TEP During Exclusive Chemo-Radiotherapy (CRT) in Patients With Oesophageal Carcinoma Cancer on the One-Year Survival (RTEP3)
Brief Title: Predictive Value of Pet Scan With Fdg Performed During Irradiation in Patients Treated for Oesaphagus Carcinoma
Acronym: RTEP3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Other Study IDs: CHB08-02
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2011-03

CONDITIONS: Oesophageal Cancer
Keywords: Positron-Emission Tomography; PET Scan; FDG; oesophageal cancer; chemo-Radiation Oncology; SUV
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The poor prognosis in the early-stage of oesophageal carcinoma cancer is due to potential worsening of the disease (local relapse, metastasis), to insufficient efficacy and toxicity of actual treatments.

FDG-PET is a medical imaging modality allowing the quantification of the tumour glucose consumption. Then, this exam is used for pathology staging, target volume definition for RT, and treatment efficiency few months after CRT. Our assumption is that an FDG-PET exam during the course of CRT might be predictive of the treatment efficiency few months later.

In this study, we propose to perform 4 FDG-PET: first "PET1" before chemo-radiotherapy, second "PET2" during the chemo-radiotherapy (see RTEP1), third and fourth "PET3" "PET4" 3month and 12 month after the end of radiotherapy.

We will investigate the performances of FDG-PET performed during CRT for the prediction of the one-year patient heath outcome. If the predictive value of TEP2 is confirmed, we would be able to optimize the planning treatment during the course of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Carcinoma épidermoïde of the oesophagus histologically proved, UICC Stage II B, III or IVa (TNM on 2002)
* Decision of treatment by radio concomitant chemotherapy (radiotherapy in classic spreading of 50Gy associated with a platinum chemotherapy.

Exclusion Criteria:

* Presence of a second evolutionary cancer in the previous three years
* index of performance OMS > 2
* Patients badly balanced diabetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed patients a carcinoma of the oesophagus histologiquement proved
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-05; Primary Completion 2013-03 (Estimated); Study Completion 2014-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: VERA Pierre, MD phD, Principal Investigator — CHBecquerel; MICHEL Pierre, MD phD, Principal Investigator — CHRU Rouen
Locations (1):
- CLCC H.Becquerel, Rouen, Haute Normandie, France

REFERENCES:
- [Derived] Nkhali L, Thureau S, Edet-Sanson A, Doyeux K, Benyoucef A, Gardin I, Michel P, Vera P, Dubray B. FDG-PET/CT during concomitant chemo radiotherapy for esophageal cancer: Reducing target volumes to deliver higher radiotherapy doses. Acta Oncol. 2015 Jun;54(6):909-15. doi: 10.3109/0284186X.2014.973062. Epub 2014 Nov 24. PMID 25417733
- [Derived] Palie O, Michel P, Menard JF, Rousseau C, Rio E, Bridji B, Benyoucef A, Meyer ME, Jalali K, Bardet S, M'vondo CM, Olivier P, Faure G, Itti E, Diana C, Houzard C, Mornex F, Di Fiore F, Vera P. The predictive value of treatment response using FDG PET performed on day 21 of chemoradiotherapy in patients with oesophageal squamous cell carcinoma. A prospective, multicentre study (RTEP3). Eur J Nucl Med Mol Imaging. 2013 Sep;40(9):1345-55. doi: 10.1007/s00259-013-2450-7. Epub 2013 May 29. PMID 23715903